CLINICAL TRIAL: NCT01925768
Title: A Phase 3b, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy and Safety of Apremilast (CC-10004) Monotherapy in Subjects With Active Psoriatic Arthritis
Brief Title: Safety and Efficacy Study of Apremilast to Treat Psoriatic Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-10004-PSA-006
Record Dates: First submitted 2013-08-15; First posted 2013-08-20 (Estimated); Results first posted 2016-06-13 (Estimated); Last update posted 2020-05-12 (Actual); Status verified 2020-04

CONDITIONS: Psoriatic Arthritis
Keywords: Apremilast, Psoriatic Arthritis, PDE4 inhibitor
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apremilast 30 mg (Experimental): 30 mg Apremilast tablets administered twice daily (BID) for 24 weeks during the double-blind placebo-controlled phase; followed by 30 mg Apremilast BID for 28 weeks of active treatment phase (up to the 52 week visit); original treatment assignments remain blinded until all participants have completed their 52 week visit or have discontinued. After the Wk 52 visit, all participants in the extension phase will continue to receive treatment with apremilast 30 mg BID until the end of the study (ie, up to Week 104 visit) or until early discontinuation from the trial.
  Interventions: Drug: Apremilast 30 mg
- Placebo (Placebo Comparator): Oral placebo BID during the placebo controlled phase weeks 0 to 24; placebo treated participants whose improvement is <10% in both swollen and tender joint counts at Week 16 are eligible for early escape (based on the measure of clinical benefit from their current treatment as evidenced by improvement (or lack of improvement) in 1) the physician (evaluator's) global assessment (EGA), 2) patients pain (pain NRS), 3) the patient global assessments (PGA), and 4) the health assessment questionnaire disability index (HAQ-DI); Placebo-treated patients who early escape are transitioned to apremilast 30 mg PO BID during the active treatment phase up to their Week 52 visit; all those who complete the 52-week treatment phase will enter an open-label extension phase for an additional 52 weeks or until early discontinuation from the trial.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apremilast 30 mg — 30mg of Apremilast will be orally administered twice daily for 104 weeks
  Other Names: Otezla; CC-10004
  Arms: Apremilast 30 mg
Drug: Placebo — Identically appearing Placebo tablets will be orally administered twice daily for up to 24 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether apremilast is safe and effective for treating patients with psoriatic arthritis.

DETAILED DESCRIPTION:
This is a Phase 3b, multicenter, randomized, double-blind, placebo-controlled, parallel-group study to evaluate the efficacy and safety of apremilast monotherapy in subjects with active psoriatic arthritis.

Approximately 214 subjects will be randomized in a 1:1 ratio to either apremilast 30 mg BID (twice a day) or identically-appearing placebo, with approximately 107 subjects per treatment group.

This is a 113-week study. The subjects will spend 24 weeks in the double-blind, placebo-controlled treatment phase, followed by 28 weeks of active treatment phase (ie, up to Week 52 visit). The original treatment assignments (apremilast 30 mg BID (twice a day) or placebo) will remain blinded until all subjects have completed their Week 52 visit (or have discontinued). After the Week 52 visit, all subjects in the extension phase will continue to receive treatment with apremilast 30 mg BID (twice a day) until the end of the study (ie, up to Week 104 visit) or until early discontinuation from the trial.

The study will consist of 5 phases:

1. Screening Phase - up to 5 weeks
2. Randomized, Placebo-controlled, Double Blind Treatment Phase - Weeks 0 to 24
3. Active Treatment Phase - Week 24 to Week 52
4. Open-label Extension Phase - Week 52 to Week 104
5. Post-treatment Observational Follow-up Phase

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, 18 years and older at time of consent.
2. Must understand and voluntarily sign an informed consent document prior to any study related assessments/procedures being conducted.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Have a documented diagnosis of psoriatic arthritis (by any criteria) of at least 3 months' duration
5. Meet the classification criteria for psoriatic arthritis (CASPAR) at the time of screening.
6. Have at least 3 swollen AND at least 3 tender joints.
7. Must have high sensitivity C-Reactive Protein (hs-CRP) of at least 0.5 mg/dL at screening and at baseline.
8. Must be receiving treatment on an outpatient basis.
9. Must be tumor necrosis factor (TNF) blocker naive and other Biologic naïve for dermatologic and rheumatic conditions
10. Subjects taking disease modifying anti-rheumatoid drugs (DMARDs), with the exception of cyclosporine and leflunomide (see 7.3. Exclusion Criteria 20, 21), do not require a washout, however, they must discontinue the DMARD treatment at least one day prior to their baseline visit (ie, Visit 2, Day 0)
11. Subjects who have been previously treated with leflunomide will require a 12-week washout or treatment with the cholestyramine, per leflunomide prescribing label (ie. 8 g cholestyramine 3 times daily for 11 days.
12. Subjects who have been previously treated with cyclosporine will require a 4-week washout prior to randomization to participate in the study
13. If taking oral corticosteroids, must be on a stable dose of prednisone less than or equal to 10 mg/day or equivalent for at least 30 days prior to baseline visit (ie, Day 0)
14. If taking nonsteroidal anti-inflammatory drugs (NSAIDs) or narcotic analgesics, must be on stable dose for at least 30 days prior to baseline visit (ie, Day 0) and until they have completed the Week 24 study visit.
15. Must meet the following laboratory criteria:

    * White blood cell count greater than 3000/mm^3 (greater than 3.0 X 10^9/L) and less than 14,000/mm^3 (less than 14 X 10^9/L)
    * Platelet count at least 100,000/mm^3 (at least 100 X 10^9/L)
    * Serum creatinine less than or equal to 1.5 mg/dL (less than or equal to 132.6 μmol/L)
    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to twice upper limit of normal (ULN). If initial test shows ALT or AST greater than 2 times the ULN, one repeat test is allowed during the screening period.
    * Total bilirubin less than or equal to 2 mg/dL (less than or equal to 34 μmol/L) or Albumin greater than LLN. If initial test result is greater than 2 mg/dL, one repeat test is allowed during the screening period.
    * Hemoglobin at least 9 g/dL (at least 5.6 mmol/L)
    * Hemoglobin A1c less than or equal to 9.0%
16. All females of childbearing potential (FCBP) must use one of the approved contraceptive options as described below while on investigational product and for at least 28 days after administration of the last dose of the investigational product.

    At the time of study entry, and at any time during the study when a female subject of childbearing potential's contraceptive measures or ability to become pregnant changes, the investigator will educate the subject regarding contraception options and the correct and consistent use of effective contraceptive methods in order to successfully prevent pregnancy.

    Females of childbearing potential must have a negative pregnancy test at Screening and Baseline. All FCBP subjects who engage in activity in which conception is possible must use one of the approved contraceptive options described below:

    Option 1: Any one of the following highly effective methods: hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation; or partner's vasectomy; OR Option 2: Male or female condom (latex condom or non latex condom NOT made out of natural [animal] membrane [for example, polyurethane]; PLUS one additional barrier method: (a) diaphragm with spermicide; (b) cervical cap with spermicide; or (c) contraceptive sponge with spermicide.
17. Male subjects (including those who have had a vasectomy) who engage in activity in which conception is possible must use barrier contraception (male latex condom or nonlatex condom NOT made out of natural [animal] membrane [for example, polyurethane]) while on investigational product and for at least 28 days after the last dose of investigational product.

Exclusion Criteria:

1. History of clinically significant (as determined by the investigator) cardiac, endocrine, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic disease, or other major uncontrolled disease.
2. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
3. Clinically significant abnormality on a 12-lead electrocardiogram (ECG) at Screening.
4. Pregnant or breast feeding.
5. History of allergy to any component of the investigational product.
6. Hepatitis B surface antigen positive at screening.
7. Hepatitis C antibody positive at screening.
8. History of positive human immunodeficiency virus (HIV), or congenital or acquired immunodeficiency (eg, Common Variable Immunodeficiency Disease).
9. Active tuberculosis or a history of incompletely treated tuberculosis.
10. Clinically significant abnormality based upon chest radiograph with at least posterior-anterior (PA) view (the radiograph must be taken within 12 weeks prior to Screening or during the Screening visit). An additional lateral view is strongly recommended but not required.
11. Active substance abuse or a history of substance abuse within 6 months prior to Screening.
12. Bacterial infections requiring treatment with oral or injectable antibiotics, or significant viral or fungal infections, within 4 weeks of Screening. Any treatment for such infections must have been completed and the infection cured, at least 4 weeks prior to Screening.
13. Malignancy or history of malignancy, except for:

    1. treated [ie, cured] basal cell or squamous cell in situ skin carcinomas;
    2. treated [ie, cured] cervical intraepithelial neoplasia [CIN] or carcinoma in situ of the cervix with no evidence of recurrence within the previous 5 years.
14. Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months following randomization.
15. Erythrodermic, guttate, or generalized pustular psoriasis at randomization.
16. Rheumatic autoimmune disease other than PsA, including, but not limited to: systemic lupus erythematosis (SLE), mixed connective tissue disease (MCTD), scleroderma, polymyositis, or fibromyalgia.
17. Functional Class IV, as defined by the American College of Rheumatology (ACR) Classification of Functional Status in Rheumatoid Arthritis.
18. Prior history of or current inflammatory joint disease other than PsA (eg, gout, reactive arthritis, rheumatoid arthritis (RA), ankylosing spondylitis, Lyme disease).
19. Prior treatment with more than one non-biologic DMARD
20. Use of the following systemic therapy(ies) within 4 weeks of randomization: cyclosporine or other calcineurin inhibitors, corticosteroids exceeding 10 mg daily prednisone equivalent, as well as other oral agents such as retinoids, mycophenolate, thioguanine, hydroxyurea, sirolimus, tacrolimus.
21. Use of leflunomide within 12 weeks of randomization, unless subject has taken cholestyramine, 8g TID (three times a day) x 11 days after stopping leflunomide.
22. Previous treatment with biologic agents for rheumatic diseases such as, but not limited to: adalimumab, abatacept, canakinumab, etanercept, golimumab, infliximab, rilonacept, certolizumab pegol, or tocilizumab.
23. Previous treatment with biologic agents for dermatologic diseases such as alefacept, anti-TNFs (eg etanercept, adalinumab) or ustekinumab.
24. Previous treatment with tofacitinib, Anti IL-17 agents or secukinumab
25. Previous treatment with any cell depleting therapies, including investigational agents (eg, rituximab, alemtuzumab, ocrelizumab, alemtuzumab, anti-CD4, anti-CD5, anti-CD3, anti-CD19, and anti-CD20).
26. Treatment with intravenous gamma globulin, plasmapheresis, or Prosorba® column
27. Any previous treatment with alkylating agents such as cyclophosphamide or chlorambucil, or with total lymphoid irradiation.
28. Prior treatment with any non-biologic DMARDS other than methotrexate, sulfasalazine, chloroquine, hydroxychloroquine, azathioprine, fumeric acid esters, cyclosporine, or leflunomide
29. Prior treatment with apremilast, or participation in a clinical study, involving apremilast
30. Use of any investigational drug within 4 weeks of randomization, or 5 pharmacokinetic/ pharmacodynamic half lives, if known (whichever is longer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2013-09-04 (Actual); Primary Completion 2015-02-25 (Actual); Study Completion 2016-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (71):
- United States (24):
  - Achieve Clinical Research LLC, Birmingham, Alabama
  - Desert Medical Advances, Palm Desert, California
  - Bay Area Arthritis and Osteoporosis, Brandon, Florida
  - Health Point Medical Group, Brandon, Florida
  - Palmetto Medical Research, Hialeah, Florida
  - Jeffrey Alper MD Research, Naples, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - University of South Florida, Tampa, Florida
  - Coeur D'Alene Arthritis Clinic, Coeur d'Alene, Idaho
  - Rockford Orthopedic Associates, LLC, Rockford, Illinois
  - Advanced Rheumatology, Lansing, Michigan
  - Research West Incorporated, Kalispell, Montana
  - Heartland Clinical Research, Inc., Omaha, Nebraska
  - Physicians East, Greenville, North Carolina
  - Piedmont Medical Research Associates Inc, Winston-Salem, North Carolina
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - West Tennessee Research Institute, Jackson, Tennessee
  - Ramesh C Gupta MD, Memphis, Tennessee
  - Austin Regional Clinic, Austin, Texas
  - Baylor Research Institute, Dallas, Texas
  - Houston Medical Research, Houston, Texas
  - Arthritis and Osteoporosis Associates LLP, Lubbock, Texas
  - University of Utah, Salt Lake City, Utah
  - Mountain State Clinical Research, Clarksburg, West Virginia
- Australia (7):
  - Colin Bayliss Research and Teaching Unit, Victoria Park, Western Australia
  - Eastern Health Clinical School, Box Hill
  - Royal Prince Alfred Hospital, Camperdown
  - Menzies Centre for Population Health Research, Hobart
  - Optimus Clinical Research Pty. Ltd, Kogarah
  - Coastal Joint Care, Maroochydore
  - Westmead Cancer Care Center, Westmead, NSW
- Canada (9):
  - Manna Research, Vancouver, British Columbia
  - Manitoba Clinic, Winnipeg, Manitoba
  - Karma Clinical Trials, St. John's, Newfoundland and Labrador
  - Nexus Clinical Research, St. John's, Newfoundland and Labrador
  - MAC Research Incorporated, Hamilton, Ontario
  - Arthur Karasik Private Practice, Toronto, Ontario
  - Manna Research, Toronto, Ontario
  - Jude Rodrigues Private Practice, Windsor, Ontario
  - CHUL du CHU de Quebec, Québec
- Czechia (4):
  - Revmatologicky ustav, Prague
  - Revmatologicka Ambulance, Prague
  - Revmatologicka Ambulance, Sokolov
  - PV - MEDICAL, s.r.o., Zlín
- Estonia (3):
  - Innomedica Medical and Research Centre, Tallinn
  - East Tallinn Central Hospital, Tallinn
  - Clinical Research Centre Ltd, Tartu
- Hungary (4):
  - Qualiclinic kft, Budapest
  - Debreceni Egyetem Orvos- es Egeszsegtudomanyi Centrum, Debrecen
  - MAV Korhaz es Rendelointezet Szolnok, Szolnok
  - Veszprém Megyei Önkormányzat Csolnoky Ferenc Kórház-Rendelöintézet, Veszprém
- New Zealand (3):
  - Waikato hospital, Hamilton
  - Middlemore Clinical Trials, Manukau
  - Timaru Hospital, Timaru
- Romania (4):
  - Sf. Maria Clinical Hospital, Bucharest
  - Emergency County Clinical Hospital, Cluj-Napoca
  - Sf Apostol Andrei Emergency Clinical County Hospital, Galati
  - SC Covamed SRL, Sfantu Gheorghe, Covasna
- Russia (4):
  - Research Medical Complex Vashe Zdorovie, Kazan'
  - Penza Regional Clinical Hospital n.a. N.N. Burdenko, Penza
  - Departmental Hospital at Smolensk Station RZhD JSC, Smolensk
  - Yaroslavl Regional Clinical Hospital, Yaroslavl
- Spain (9):
  - Hospital Universitario a Coruna, A Coruña
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona, Hospitalet de Llobregat
  - Hospital de Basurto-Osakidetza, Bilbao
  - Hospital Universitario La Paz, Madrid
  - Hospital General Carlos Haya, Málaga
  - Corporacion Sanitaria Parc Tauli, Sabadell
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Nash P, Ohson K, Walsh J, Delev N, Nguyen D, Teng L, Gomez-Reino JJ, Aelion JA; ACTIVE investigators. Early and sustained efficacy with apremilast monotherapy in biological-naive patients with psoriatic arthritis: a phase IIIB, randomised controlled trial (ACTIVE). Ann Rheum Dis. 2018 May;77(5):690-698. doi: 10.1136/annrheumdis-2017-211568. Epub 2018 Jan 17. PMID 29343507
- [Derived] Mease PJ, Hatemi G, Paris M, Cheng S, Maes P, Zhang W, Shi R, Flower A, Picard H, Stein Gold L. Apremilast Long-Term Safety Up to 5 Years from 15 Pooled Randomized, Placebo-Controlled Studies of Psoriasis, Psoriatic Arthritis, and Behcet's Syndrome. Am J Clin Dermatol. 2023 Sep;24(5):809-820. doi: 10.1007/s40257-023-00783-7. Epub 2023 Jun 14. PMID 37316690

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted of a 24-week randomized, double-blind, placebo-controlled treatment phase, followed by a 28-week active treatment phase and a 52-week open-label extension phase, for an overall study duration of 113 weeks. 219 subjects were enrolled from 59 centers across 10 countries.
Pre-assignment Details: Randomized participants were stratified by their baseline prednisone use (yes or no) and by their previous disease modifying antirheumatic drug (DMARD) use (excluding biologics). Participants were allowed to take non-steroidal anti-inflammatory agents and/or low dose corticosteroids during the study.
Groups:
- Placebo/Apremilast (PBO): Participants were randomized to placebo tablets twice daily (BID) during the double-blind, 24-week placebo-controlled phase. Those whose improvement was less than 10% in both swollen and tender joint counts at Week 16 were eligible for early escape (EE), at the discretion of the investigator and transitioned onto apremilast 30 mg BID in a blinded fashion. Those who had a 10% or more improvement in either swollen or tender joint counts at Week 16 were not eligible for early escape. Participants who completed the double-blind, 24-week treatment phase entered into the blinded, active treatment phase for an additional 28 weeks (Week 24 to Week 52) and continued receiving Apremilast 30 mg tablets BID. Participants who completed the active treatment phase entered into the open-label extension phase for an additional year (Week 52 to Week 104) continuing to receive apremilast 30 mg tablets BID until the end of the study (up to Week 104 visit) or until early discontinuation.
- Apremilast (APR): Participants were randomized to apremilast 30 mg tablets BID during the double-blind, 24-week placebo-controlled phase. Those whose improvement was less than 10% in both swollen and tender joint counts at Week 16 were eligible for early escape, at the discretion of the investigator and continued receiving apremilast 30 mg BID in a blinded fashion. Those who had a 10% or more improvement in either swollen or tender joint counts at Week 16 were not eligible for early escape. Participants who completed the double-blind 24-week treatment phase entered into the blinded active treatment phase for an additional 28 weeks (Week 24 to Week 52) and continued receiving Apremilast 30 mg tablets BID. All participants who completed the 52-week treatment phase entered into the open-label extension phase (Week 52 to Week 104) for an additional year continuing to receive apremilast 30 mg tablets BID until the end of the study (up to Week 104 visit) or until early discontinuation.
Period: Placebo-controlled Phase (Week 0 - 24)
Arm/Group | Placebo/Apremilast (PBO) | Apremilast (APR)
Started | 109 | 110
Received Treatment | 109 | 109
Completed Week 16 | 101 | 91
Escaped Early (EE) | 35 | 13
Completed | 98 (3 participants who completed Week 24 did not enter the active treatment phase) | 87 (2 participants who completed Week 24 did not enter the active treatment phase)
Not Completed | 11 | 23
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 1 | 2
Not completed — Adverse Event | 5 | 10
Not completed — Lack of Efficacy | 3 | 6
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Non-compliance with study drug | 0 | 1
Period: ActiveTreatment/Extension (Weeks 24-104)
Arm/Group | Placebo/Apremilast (PBO) | Apremilast (APR)
Started | 95 | 85
Completed | 75 | 67 (Completed Apremilast treatment at Week 104)
Not Completed | 20 | 18
Not completed — Lack of Efficacy | 6 | 6
Not completed — Withdrawal by Subject | 7 | 9
Not completed — Lost to Follow-up | 2 | 1
Not completed — Death | 0 | 1
Not completed — Adverse Event | 5 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set consisting of all participants who were randomized as specified in the protocol.
Groups:
- Placebo (PBO): Participants randomized to placebo tablets BID during the blinded, 24-week placebo-controlled phase. Participants whose improvement was less than 10% in both swollen and tender joint counts at Week 16 were eligible for early escape (EE), at the discretion of the investigator were transitioned onto apremilast 30 mg tablets BID in a blinded fashion. Those who had a 10% or more improvement in either swollen or tender joint counts at Week 16 were not eligible for early escape.
- Apremilast (APR) 30 mg: Participants randomized to apremilast 30 mg tablets BID during the blinded, 24-week placebo-controlled phase. Participants whose improvement was less than 10% in both swollen and tender joint counts at Week 16 were eligible for EE, at the discretion of the investigator and continued receiving apremilast 30 mg BID in a blinded fashion. Those who had a 10% or more improvement in either swollen or tender joint counts at Week 16 were not eligible for early escape.
- Total: Total of all reporting groups
Arm/Group | Placebo (PBO) | Apremilast (APR) 30 mg | Total
Number analyzed (Participants) | 109 | 110 | 219
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (13.75) | 50.7 (12.22) | 49.3 (13.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 58 | 123
  Male | 44 | 52 | 96
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 0 | 1
  White | 105 | 109 | 214
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Duration of Psoriatic Arthritis [Mean (Standard Deviation); unit: years] — Duration of Psoriatic Arthritis is reported as the time since diagnosis
  years | 3.59 (5.497) | 4.04 (4.482) | 3.82 (5.007)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved an American College of Rheumatology 20% (ACR20) Response at Week 16
Description: Percentage of participants with an American College of Rheumatology 20% (ACR20) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met:
  * ≥ 20% improvement in 78 tender joint count;
  * ≥ 20% improvement in 76 swollen joint count; and
  * ≥ 20% improvement in at least 3 of the 5 following parameters:
    * Patient's self-assessment of pain (measured on a 0 to 10 unit numeric rating scale [NRS]);
    * Patient's global self-assessment of disease activity (measured on a 0 to 10 unit NRS);
    * Physician's global assessment of disease activity (measured on a 0 to 10 unit NRS);
    * Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI]);
    * C-Reactive Protein (CRP) Those who withdrew early or who did not have sufficient data at Week 16 were counted as non-responders.
Time Frame: Baseline and Week 16
Population: Full Analysis Set (FAS) population consisting of all participants randomized as specified in the protocol.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (PBO) | Apremilast (APR) 30 mg
Number analyzed (Participants) | 109 | 110
percentage of participants | 20.2 | 38.2
Statistical Analysis 1: Comparison: Placebo (PBO) vs Apremilast (APR) 30 mg; Test type: Superiority or Other; p = 0.0040, Cochran-Mantel-Haenszel — Two-sided p-value is based on the Cochran-Mantel-Haenszel test adjusting for previous DMARD use and baseline Oral Corticosteroids (Prednisone or equivalent) use; Adjusted Difference = 17.7, 95% CI 2-sided [6.2 to 29.3] — Adjusted difference in proportions is the weighted average of the treatment differences across 4 strata by the 2 stratification factors: previous DMARD use and baseline Corticosteroids use using CMH weights. The CI is based on a normal approximation

2. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) at Week 24
Description: HAQ-DI is a patient-reported questionnaire consisting of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and usual activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task are summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. A higher score indicates worse physical functioning, and a negative change from baseline indicates improvement.
Time Frame: Baseline and Week 24
Population: Full analysis set; Participants with a baseline and at least 1 postbaseline value during the placebo-controlled phase were included in the analysis (mixed effects model for repeated measure [MMRM])
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (PBO) | Apremilast (APR) 30 mg
Number analyzed (Participants) | 109 | 109
units on a scale | -0.169 (0.0581) | -0.273 (0.0572)
Statistical Analysis 1: Comparison: Placebo (PBO) vs Apremilast (APR) 30 mg; Test type: Superiority or Other; p = 0.1677, Mixed Models Analysis; Those with a baseline and at least 1 postbaseline value at the PBO controlled phase were counted with mixed effects model for repeated measure (MMRM); LS Mean Difference = -0.103, 95% CI 2-sided [-0.251 to 0.044] — The LS mean (SE) and 2-sided p-value were based on a MMRM analysis for change from baseline, with treatment group, time, treatment-by-time interaction, and previous DMARD and baseline corticosteroids used as factors and baseline value as a covariate

3. Secondary Outcome: Percentage of Participants Who Achieved an American College of Rheumatology 20% (ACR20) at Week 24
Description: as for outcome 1
Time Frame: Baseline and Week 24
Population: FAS population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (PBO) | Apremilast (APR) 30 mg
Number analyzed (Participants) | 109 | 110
percentage of participants | 24.8 | 43.6
Statistical Analysis 1: Comparison: Placebo (PBO) vs Apremilast (APR) 30 mg; Test type: Superiority or Other; p = 0.0040, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Those who withdrew early or who did not have sufficient data at Week 16 were counted as non-responders; Adjusted Difference = 18.5, 95% CI 2-sided [6.3 to 30.6] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline in the 28-Joint Disease Activity Score Using C-reactive Protein as the Acute-Phase Reactant (DAS28 [CRP]) at Week 24
Description: The DAS28 measures the severity of disease at a specific time and is derived from the following variables:
  * 28 tender joint count
  * 28 swollen joint count, which do not include the DIP joints, the hip joint, or the joints below the knee;
  * C-reactive protein (CRP)
  * Patient's global assessment of disease activity. DAS28 (CRP) scores range from 0 to 9.4. A DAS28 score higher than 5.1 indicates high disease activity, a DAS28 score less than 3.2 indicates low disease activity, and a DAS28 score less than 2.6 indicates clinical remission. A higher value indicates higher disease activity, and a negative change from baseline indicates improvement.
Time Frame: Baseline and Week 24
Population: Full analysis set; Participants with a baseline value and at least one post-baseline value (after exclusion of data for early escaped participants) during the placebo-controlled phase are included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (PBO) | Apremilast (APR) 30 mg
Number analyzed (Participants) | 108 | 109
units on a scale | -0.76 (0.140) | -1.26 (0.138)
Statistical Analysis 1: Comparison: Placebo (PBO) vs Apremilast (APR) 30 mg; Test type: Superiority or Other; p = 0.0051, Mixed Models Analysis; LS Mean Difference = -0.50, 95% CI 2-sided [-0.85 to -0.15] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Change From Baseline in the Medical Outcomes Short Form Health Survey (SF-36) V2 Physical Function Domain Score at Week 24
Description: The Medical Outcome Study Short Form 36-Item Health Survey, Version 2 (SF-36) is a self-administered instrument that measures the impact of disease on overall quality of life and consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health). Norm-based scores were used in analyses, calibrated so that 50 is the average score and the standard deviation equals 10. Higher scores indicate a higher level of functioning. The physical functioning domain assesses limitations in physical activities because of health problems. A positive change from baseline score indicates an improvement.
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (PBO) | Apremilast (APR) 30 mg
Number analyzed (Participants) | 106 | 107
units on a scale | 1.26 (0.908) | 3.94 (0.888)
Statistical Analysis 1: Comparison: Placebo (PBO) vs Apremilast (APR) 30 mg; Test type: Superiority or Other; p = 0.0167, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = 2.68, 95% CI 2-sided [0.49 to 4.88] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Change From Baseline in the 36-item SF-36 Physical Component Summary Score at Week 24
Description: The SF-36 (v 2.0) is a self-administered instrument that measures the impact of disease on overall quality of life and consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health). The physical component summary (PCS) score includes the physical functioning, role physical, bodily pain, and general health domains. Minimum clinically important difference (MCID) for the scale scores, as well as the PCS and MCS, is defined as a 2.5-point improvement (increase) from baseline. The summary scores range from 0 to 100, with lower scores reflecting more disability, and higher scores reflecting less disability and better health. The 8 domains are regrouped into the PCS and MCS scores.
Time Frame: Baseline and Week 24
Population: Full analysis set. Subjects with a baseline value and at least one post-baseline value (after exclusion of data for early escaped subjects) during the placebo-controlled phase are included in the MMRM model.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (PBO) | Apremilast (APR) 30 mg
Number analyzed (Participants) | 106 | 106
units on a scale | 1.60 (0.959) | 5.00 (0.949)
Statistical Analysis 1: Comparison: Placebo (PBO) vs Apremilast (APR) 30 mg; 2-sided 95% CI for the difference in LS mean; Test type: Superiority or Other; p = 0.0039, Mixed Models Analysis — Based on an MMRM model for the change from baseline, with treatment group, time, treatment-by-time interaction, and previous DMARD use and baseline Oral Corticosteroids use as factors and the baseline value as a covariate; LS Mean Difference = 3.40, 95% CI 2-sided [1.10 to 5.70]

7. Secondary Outcome: Change From Baseline in the Duration of Morning Stiffness at Week 24
Description: Morning stiffness was the participant's assessment of how long their morning stiffness lasted after first waking up in the morning, on average, during the previous week. A higher value indicates longer duration, and a negative change from baseline indicates improvement.
Time Frame: Baseline and Week 24
Population: Full Analysis Set; Analysis includes participants with a baseline and at least one post-baseline value; last observation carried forward (LOCF) imputation was used
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo (PBO) | Apremilast (APR) 30 mg
Number analyzed (Participants) | 109 | 109
minutes | 21.9 (137.11) [-460 to -879] | -5.7 (83.41) [-175 to -679]
Statistical Analysis 1: Comparison: Placebo (PBO) vs Apremilast (APR) 30 mg; Test type: Superiority or Other; p = 0.012, Sign test; p-value based on distribution free signed rank test; Mean Difference (Final Values) = -10.0, 95% CI 2-sided [-21.5 to 10.2]

8. Secondary Outcome: Percentage of Participants With Improved Change in Severity of Morning Stiffness at Week 24
Description: Morning stiffness severity was the participant's assessment of how severe their morning stiffness was after first waking up in the morning, on average, during the previous week. The severity was recorded as none, mild, moderate, moderately severe, or very severe. The response of no improvement includes subjects who had no change or worsened. Improvement is defined as the change from baseline of a more severe assessment to less severe assessment.
Time Frame: Baseline and Week 24
Population: Full Analysis Set; Participants who withdrew early or who did not have sufficient data at Week 24 were counted as non-responders
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (PBO) | Apremilast (APR)
Number analyzed (Participants) | 109 | 110
percentage of participants | 20.2 | 40.0
Statistical Analysis 1: Comparison: Placebo (PBO) vs Apremilast (APR); Test type: Superiority or Other; p = 0.0016, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted Difference = 19.7, 95% CI 2-sided [8.0 to 31.3] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) at Week 16
Description: as for outcome 2
Time Frame: Baseline and Week 16
Population: Full analysis set; participants with a baseline value and at least 1 postbaseline value during the placebo-controlled phase were included in the mixed effects model for repeated measures (MRMM).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (PBO) | Apremilast (APR) 30 mg
Number analyzed (Participants) | 109 | 109
units on a scale | -0.055 (0.0513) | -0.205 (0.0523)
Statistical Analysis 1: Comparison: Placebo (PBO) vs Apremilast (APR) 30 mg; Test type: Superiority or Other; p = 0.0229, Mixed Models Analysis; LS Mean Difference = -0.150, 95% CI 2-sided [-0.279 to -0.021] — [estimate comment as in outcome 2, analysis 1]

10. Secondary Outcome: Change From Baseline in the Disease Activity Score DAS28 (CRP) at Week 16
Description: The DAS28 measures the severity of disease at a specific time and is derived from the following variables:
  * 28 tender joint count
  * 28 swollen joint count, which do not include the DIP joints, the hip joint, or the joints below the knee;
  * C-reactive protein (CRP)
  * Patient's global assessment of disease activity. DAS28 (CRP) scores range from 0 to 9.4. A DAS28 score higher than 5.1 indicates high disease activity, a DAS28 score less than 3.2 indicates low disease activity, and a DAS28 score less than 2.6 indicates clinical remission. A negative change from baseline indicates improvement.
Time Frame: Baseline and Week 16
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (PBO) | Apremilast (APR) 30 mg
Number analyzed (Participants) | 108 | 109
units on a scale | -0.39 (0.129) | -1.07 (0.133)
Statistical Analysis 1: Comparison: Placebo (PBO) vs Apremilast (APR) 30 mg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -0.68, 95% CI 2-sided [-1.00 to -0.35] — [estimate comment as in outcome 2, analysis 1]

11. Secondary Outcome: Change From Baseline in 36-item Short Form Health Survey (SF-36) V 2 Physical Functioning Domain at Week 16
Description: The SF-36 (v 2.0) is a self-administered instrument that measures the impact of disease on overall quality of life and consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health). Norm-based scores were used in analyses, calibrated so that 50 is the average score and the standard deviation equals 10. Higher scores indicate a higher level of functioning. The physical functioning domain assesses limitations in physical activities because of health problems. A positive change from Baseline score indicates an improvement.
Time Frame: Baseline and Week 16
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (PBO) | Apremilast (APR) 30 mg
Number analyzed (Participants) | 106 | 107
units on a scale | -1.04 (0.927) | 2.43 (0.962)
Statistical Analysis 1: Comparison: Placebo (PBO) vs Apremilast (APR) 30 mg; Test type: Superiority or Other; p = 0.0039, Mixed Models Analysis; LS Mean Difference = 3.46, 95% CI 2-sided [1.13 to 5.80] — Adjusted difference in proportions is the weighted average of the treatment differences across 4 strata by the 2 stratification factors: previous DMARD use and baseline Corticosteroids use using CMH weights

12. Secondary Outcome: Mean Change From Baseline in the Duration of Morning Stiffness at Week 16
Description: as for outcome 7
Time Frame: Baseline and Week 16
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo (PBO) | Apremilast (APR) 30 mg
Number analyzed (Participants) | 109 | 109
minutes | 21.7 (136.85) | -7.2 (60.73)
Statistical Analysis 1: Comparison: Placebo (PBO) vs Apremilast (APR) 30 mg; Test type: Superiority or Other; p = 0.0168, Stratified Van Elteren test; p-value based on stratified Van Elteren test, using 2 stratification factors: previous DMARD use and baseline Oral Corticosteroids; Hodges-Lehmann = 10.0, 95% CI 2-sided [0.0 to 20.0] — Location shift and 95% CI based on Hodges-Lehmann for between treatment median estimates

13. Secondary Outcome: Percentage of Participants Whose Severity of Morning Stiffness at Week 16 Improved From Baseline
Description: Morning stiffness severity was the participant's assessment of how severe their morning stiffness was after first waking up in the morning, on average, during the previous week. The severity was recorded as none, mild, moderate, moderately severe, or very severe. Improvement is defined as the change from baseline of a more severe assessment to less severe assessment. Full Analysis Set; Participants who discontinued early prior to Week 16 and those who did not have sufficient data for a definitive determination of response status at Week 16 were counted as non-responders.
Time Frame: Baseline and Week 16
Population: Full Analysis Set; Participants who discontinued early prior to Week 16 and those who did not have sufficient data for a definitive determination of response status at Week 16 were counted as non-responders
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (PBO) | Apremilast (APR) 30 mg
Number analyzed (Participants) | 109 | 110
percentage of participants | 25.7 | 46.4
Statistical Analysis 1: Comparison: Placebo (PBO) vs Apremilast (APR) 30 mg; Test type: Superiority or Other; p = 0.0015, Cochran-Mantel-Haenszel — 2 sided-p-value is based on the Cochran-Mantel-Haenszel test adjusting for previous DMARD use and baseline Oral Corticosteroids (Prednisone or equivalent) use; Adjusted Difference = 20.7, 95% CI 2-sided [8.5 to 32.8] — [estimate comment as in outcome 11, analysis 1]

14. Secondary Outcome: Percentage of Participants Who Achieved an American College of Rheumatology 20% (ACR20) Response at Weeks 2, 4, 6, 8, 12 and 20
Description: Percentage of participants with an American College of Rheumatology 20% (ACR20) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met:
  * ≥ 20% improvement in 78 tender joint count;
  * ≥ 20% improvement in 76 swollen joint count; and
  * ≥ 20% improvement in at least 3 of the 5 following parameters:
    * Patient's self-assessment of pain (measured on a 0 to 10 unit numeric rating scale [NRS]);
    * Patient's global self-assessment of disease activity (measured on a 0 to 10 unit NRS);
    * Physician's global assessment of disease activity (measured on a 0 to 10 unit NRS);
    * Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI]);
    * C-Reactive Protein (CRP)
Time Frame: Baseline and at Weeks 2, 4, 6, 8, 12 and 20
Population: Full analysis set; participants discontinued early prior to the visit and participants who did not have sufficient data for a definitive determination of response status for the visit were counted as nonresponders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (PBO) | Apremilast (APR) 30 mg
Number analyzed (Participants) | 109 | 110
percentage of participants
  Week 2 | 6.4 | 16.4
  Week 4 | 15.6 | 24.5
  Week 6 | 19.3 | 37.3
  Week 8 | 22.9 | 36.4
  Week 12 | 28.4 | 40.0
  Week 20 | 24.8 | 43.6
Statistical Analysis 1: Comparison: Placebo (PBO) vs Apremilast (APR) 30 mg; Week 2; 2-sided 95% CI is based on a normal approximation to the weighted average; Test type: Superiority or Other; p = 0.0252, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted Difference = 9.7, 95% CI 2-sided [1.6 to 17.7] — Adjusted difference in proportions is the weighted average of the treatment differences across 4 strata by 2 stratification factors: previous DMARD use and baseline Corticosteroids use using CMH weights
Statistical Analysis 2: Comparison: Placebo (PBO) vs Apremilast (APR) 30 mg; Week 4; 2-sided 95% CI is based on a normal approximation to the weighted average; Test type: Superiority or Other; p = 0.1121, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted Difference = 8.6, 95% CI 2-sided [-1.7 to 18.9] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 3: Comparison: Placebo (PBO) vs Apremilast (APR) 30 mg; Week 6; 2-sided 95% CI is based on a normal approximation to the weighted average; Test type: Superiority or Other; p = 0.0036, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted Difference = 17.8, 95% CI 2-sided [6.2 to 29.3] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 4: Comparison: Placebo (PBO) vs Apremilast (APR) 30 mg; Week 8; 2-sided 95% CI is based on a normal approximation to the weighted average; Test type: Superiority or Other; p = 0.0392, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted Difference = 12.7, 95% CI 2-sided [0.8 to 24.6] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 5: Comparison: Placebo (PBO) vs Apremilast (APR) 30 mg; Week 12; 2-sided 95% CI is based on a normal approximation to the weighted average; Test type: Superiority or Other; p = 0.0884, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted Difference = 11.0, 95% CI 2-sided [-1.3 to 23.2] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 6: Comparison: Placebo (PBO) vs Apremilast (APR) 30 mg; Week 20; 2-sided 95% CI is based on a normal approximation to the weighted average; Test type: Superiority or Other; p = 0.0040, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted Difference = 18.6, 95% CI 2-sided [6.5 to 30.7] — [estimate comment as in outcome 14, analysis 1]

15. Secondary Outcome: Percentage of Participants Who Achieved an American College of Rheumatology 20% (ACR20) Response at Weeks 52 and 104
Description: as for outcome 14
Time Frame: Baseline and Weeks 52 and 104
Population: Apremilast Participants as Randomized or Transitioned, which includes all participants who randomized or escaped/transitioned (at Week 16 or Week 24) to apremilast, and with available data at each time point.
Measure: Number (95% Confidence Interval); unit: percentage of partcipants
Groups:
- Placebo/Apremilast (PBO-APR): Participants initially randomized to placebo tablets BID in the 24-week place controlled phase. Participants whose improvement was less than 10% in both swollen and tender joint counts at Week 16 were eligible for early escape (EE), at the discretion of the investigator. Placebo-treated participants who required EE were transitioned to apremilast 30 mg BID in a blinded fashion and remained on their original treatment assignment.
Arm/Group | Placebo/Apremilast (PBO-APR) | Apremilast (APR)
Number analyzed (Participants) | 90 | 79
percentage of partcipants
  Week 52 | 60.0 [49.1 to 70.2] | 67.1 [55.6 to 77.3]
  Week 104: number analyzed (Participants) | 74 | 69
  Week 104 | 66.2 [54.3 to 76.8] | 59.4 [46.9 to 71.1]

16. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) at Weeks 52 and 104
Description: as for outcome 2
Time Frame: Baseline and Weeks 52 and 104
Population: Apremilast participants as randomized or transitioned; The Placebo/Apremilast 30 mg BID group includes participants initially randomized to placebo and switched to apremilast 30 mg BID at Week 16 or 24 and with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo/Apremilast (PBO-APR) | Apremilast (APR)
Number analyzed (Participants) | 91 | 80
units on a scale
  Week 52 | -0.323 (0.5759) | -0.395 (0.5297)
  Week 104: number analyzed (Participants) | 75 | 69
  Week 104 | -0.382 (0.5639) | -0.357 (0.6102)

17. Secondary Outcome: Change From Baseline in the Disease Activity Score (DAS28) at Week 52 and 104
Description: as for outcome 10
Time Frame: Baseline and Weeks 52 and 104
Population: Apremilast participants as randomized or transitioned. The Placebo/Apremilast30 mg BID group includes participants initially randomized to placebo and switched to apremilast 30 mg BID at Week 16 or 24 and with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo/Apremilast (PBO-APR) | Apremilast (APR)
Number analyzed (Participants) | 90 | 79
units on a scale
  Week 52 | -1.46 (0.985) | -1.71 (1.054)
  Week 104: number analyzed (Participants) | 73 | 69
  Week 104 | -1.62 (1.086) | -1.70 (1.305)

18. Secondary Outcome: Change From Baseline in 36-item SF-36 (V2.0) Physical Functioning Domain Score at Weeks 52 and 104
Description: as for outcome 11
Time Frame: Baseline and Weeks 52 and 104
Population: Apremilast Subjects as Randomized or Transitioned; The Placebo/30 mg BID group includes participants initially randomized to placebo and switched to apremilast 30 mg BID at Week 16 or 24and with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo/Apremilast (PBO-APR) | Apremilast (APR)
Number analyzed (Participants) | 91 | 80
units on a scale
  Week 52 | 5.11 (9.842) | 6.00 (9.990)
  Week 104: number analyzed (Participants) | 75 | 69
  Week 104 | 5.78 (9.932) | 5.95 (10.827)

19. Secondary Outcome: Change From Baseline in the Duration of Morning Stiffness at Weeks 52 and 104
Description: as for outcome 7
Time Frame: Baseline and Weeks 52 and 104
Population: Apremilast participants as randomized or transitioned; The Placebo/ Apremilast 30 mg BID group includes participants initially randomized to placebo and switched to apremilast 30 mg BID at Week 16 or 24 And with available data at each time point.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo/Apremilast (PBO-APR) | Apremilast (APR)
Number analyzed (Participants) | 91 | 80
minutes
  Week 52 | 3.3 (174.41) | -5.7 (93.62)
  Week 104: number analyzed (Participants) | 75 | 69
  Week 104 | -11.9 (165.36) | -7.0 (71.34)

20. Secondary Outcome: Percentage of Participants Whose Severity of Morning Stiffness at Week 52 and 104 Improved From Baseline
Description: Morning stiffness severity was the participant's assessment of how severe their morning stiffness was after first waking up in the morning, on average, during the previous week. The severity was recorded as none, mild, moderate, moderately severe, or very severe. Improvement is defined as the change from baseline of a more severe assessment to less severe assessment.
Time Frame: Baseline and Weeks 52 and 104
Population: Apremilast participants as randomized or transitioned. The Placebo/30 mg BID group includes subjects initially randomized to placebo and switched to apremilast 30 mg BID at Week 16 or 24 and with available data at each time point
Measure: Number; unit: percentage of participants
Arm/Group | Placebo/Apremilast (PBO-APR) | Apremilast (APR)
Number analyzed (Participants) | 91 | 80
percentage of participants
  Week 52 | 57.1 | 57.5
  Week 104: number analyzed (Participants) | 75 | 69
  Week 104 | 50.7 | 59.4

21. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE) During the 24 Week Placebo Controlled Phase
Description: A TEAE is an AE with a start date on or after the date of the first dose of Investigational Product (IP). An AE is any noxious, unintended, or untoward medical occurrence, that may appear or worsen in a participant during the course of study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the participant's health, including laboratory test values regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a preexisting condition) was considered an AE. A serious AE (SAE) is any untoward adverse event that is fatal, life-threatening, results in persistent or significant disability or incapacity, requires or prolongs existing in-patient hospitalization, is a congenital anomaly or birth defect, or a condition that may jeopardize the patient or may require intervention to prevent one of the outcomes listed above.
Time Frame: Date of first dose of study drug to Week 24; median duration of exposure during placebo controlled phase was 24.14 weeks
Population: Safety population includes all participants who were randomized and received at least one dose of IP.
Measure: Number; unit: Participants
Arm/Group | Placebo (PBO) | Apremilast (APR) 30 mg
Number analyzed (Participants) | 109 | 109
Participants
  Any TEAE | 69 | 73
  Any drug-related TEAE | 18 | 30
  Any severe TEAE | 4 | 2
  Any serious TEAE | 5 | 3
  Any serious drug-related TEAE | 0 | 0
  Any TEAE leading to study drug withdrawal | 5 | 10
  Any TEAE leading to study dose interruption | 7 | 10
  Any TEAE leading to death | 0 | 0

22. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE) During the Apremilast-Exposure Period
Description: as for outcome 21
Time Frame: Start of lst dose of IP up to week 104: Weeks 0 to104 for those initially randomized to APR 30 mg BID, Weeks 16 -104 for PBO-treated patients who EE to APR at Week 16 and from Weeks 24-104 for PBO-treated patients who transitioned to APR at Week 24
Population: APR participants as treated (AAT) population; AAT = participants who received at least 1 dose of APR at any time during the study, (those initially randomized to the APR 30 BID at Week 0, those initially randomized to placebo who entered EE and transitioned to APR at Week 16, and those initially randomized to PBO who transitioned to APR at Week 24)
Measure: Number; unit: Participants
Arm/Group | Apremilast (APR) 30 mg
Number analyzed (Participants) | 206
Participants
  Any TEAE | 157
  Any drug-related TEAE | 52
  Any severe TEAE | 8
  Any serious TEAE | 15
  Any serious drug-related TEAE | 0
  Any TEAE leading to study dose interruption | 28
  Any TEAE leading to study drug withdrawal | 17
  Any TEAE leading to death | 1

ADVERSE EVENTS:
Time Frame: AE's are reported: 1. Placebo-controlled phase (Weeks 0-24) 2. Up to 104 weeks for all participants randomized or transitioned onto apremilast at any time during the study (apremilast-exposure phase). AEs were monitored for 37 months
Description: Median duration of exposure during the placebo-controlled phase was 24.14 weeks and 81 weeks during the apremilast exposure phase.
Groups:
- Placebo-Controlled Phase: Placebo (Weeks 0-24): Participants who were randomized to placebo tablets twice daily (BID) during the double-blind, 24-week placebo-controlled phase.
- Placebo-Controlled Phase: Apremilast (Weeks 0-24): Participants who were randomized to apremilast tablets twice daily during the double-blind, 24-week placebo-controlled phase.
- APR Exposure Period: Apremilast: Participants who received apremilast any point during the course of the study, on Day 0, 16 or Day 24 and continued to receive apremilast 30 mg tablets BID up to week 104.
Arm/Group | Placebo-Controlled Phase: Placebo (Weeks 0-24) | Placebo-Controlled Phase: Apremilast (Weeks 0-24) | APR Exposure Period: Apremilast
Serious Adverse Events (participants affected / at risk) | 5/109 | 3/109 | 15/206
Other Adverse Events (participants affected / at risk) | 37/109 | 41/109 | 83/206
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-Controlled Phase: Placebo (Weeks 0-24) (N=109) | Placebo-Controlled Phase: Apremilast (Weeks 0-24) (N=109) | APR Exposure Period: Apremilast (N=206)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Cardiomyopathy alcoholic (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 2
Hypertensive heart disease (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Arthritis infective (Infections and infestations) | 0 | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 1
Spinal column injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Respiratory papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-Controlled Phase: Placebo (Weeks 0-24) (N=109) | Placebo-Controlled Phase: Apremilast (Weeks 0-24) (N=109) | APR Exposure Period: Apremilast (N=206)
Diarrhoea (Gastrointestinal disorders) | 12 | 16 | 34
Nausea (Gastrointestinal disorders) | 2 | 9 | 18
Bronchitis (Infections and infestations) | 3 | 5 | 11
Nasopharyngitis (Infections and infestations) | 7 | 9 | 17
Upper respiratory tract infection (Infections and infestations) | 11 | 5 | 17
Headache (Nervous system disorders) | 4 | 8 | 13
Hypertension (Vascular disorders) | 7 | 7 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is more than 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 days. Investigator must delete confidential information before submission or defer publication to permit patent applications